CLINICAL TRIAL: NCT03539172
Title: A Phase II Trial of Radiotherapy Concurrent With Apatinib in Advanced Soft Tissue and Bone Sarcomas of Head and Neck: the RASS Study
Brief Title: Radiotherapy Concurrent With Apatinib in Advanced Soft Tissue and Bone Sarcomas of Head and Neck--RASS Study
Acronym: RASS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018HNRT01
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Soft Tissue and Bone Tumor; Head and Neck Cancer; Sarcoma
MeSH Terms: conditions — Neoplasms, Connective and Soft Tissue; Head and Neck Neoplasms; Sarcoma | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib group (Experimental): Apatinib Mesylate administered as a daily oral treatment
  Interventions: Drug: Apatinib Mesylate

INTERVENTIONS:
Drug: Apatinib Mesylate — Apatinib Mesylate will be administered orally at 500 mg once daily from 2 weeks before the beginning of radiotherapy until the end of whole radiotherapy course

SUMMARY:
This is a non-randomized, phase II, open label study of radiotherapy concurrent with Apatinib Mesylate after surgery in patients with advanced head and neck soft tissue and bone sarcomas. The primary purpose of this study is to evaluate the efficacy and safety of Apatinib Mesylate in patients with head and neck soft tissue and bone sarcomas.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of head and neck soft tissue sarcoma (undifferentiated pleomorphic sarcoma, synovial sarcoma, alveolar soft part sarcoma, clear cell sarcoma, angiosarcoma, epithelioid hemangiosarcoma, solitary fibrous tumor and epithelioid sarcomas) or bone sarcoma (osteosarcoma/high grade bone sarcoma, Ewing sarcoma or dedifferentiated chondrosarcoma) confirmed by central pathology review.
2. Gross total resection, with Invasive cancer seen on microscopic evaluation of the resection margin, or with gross tumor residual, or surgically unresectable and/or refuse surgery.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
4. Adequate hepatic, renal, cardiac, and hematologic function.
5. Patients must provide written informed consent prior to performance of study-specific procedures and must be willing to comply with treatment and follow-up.

Exclusion Criteria:

1. Evidence of distant metastasis
2. Prior chemotherapy or anti-cancer biologic therapy for any type of cancer, or prior radiotherapy to the head and neck region
3. Other previous cancer, except for in situ cervical cancer and cutaneous basal cell carcinoma
4. Pregnant or breast-feeding females, or females and males of childbearing potential not taking adequate contraceptive measures
5. Presence of an uncontrolled concomitant illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
6. Suffered from grade II or above myocardial ischemia or myocardial infarction, uncontrolled arrhythmias (including QT interval male ≥ 450 ms, female ≥ 470 ms). Grade III-IV cardiac insufficiency according to New York Heart Association (NYHA) criteria or echocardiography check: left ventricular ejection fraction (LVEF)<50%
7. Patients who have had prior allergic reaction to Apatinib

Ages: 10 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | 2 year
  To determine 2 year PFS of Apatinib Mesylate when administered as monotherapy in patients with metastatic adenoid cystic carcinoma

SECONDARY OUTCOMES:
Overall survival rate | 2 year
  from date of enrollment until date of first death from any cause, assessed up to 2 years
Number of participants with treatment-related adverse events as assessed by CTCAE v3.0 | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai ninth people's hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided